CLINICAL TRIAL: NCT03719326
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of Immunotherapy Combinations in Participants With Breast or Gynecologic Malignancies
Brief Title: A Study to Evaluate Safety/Tolerability of Immunotherapy Combinations in Participants With Triple-Negative Breast Cancer or Gynecologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-2 (AB928CSP0002)
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Ovarian Cancer
Keywords: Triple Negative Breast Cancer; TNBC; Ovarian Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Ovarian Neoplasms | interventions — IPI-549; liposomal doxorubicin; Taxes

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation-Arm A (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period.
  Interventions: Drug: Etrumadenant; Drug: Pegylated liposomal doxorubicin (PLD)
- Dose Escalation-Arm B (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period.
  Interventions: Drug: Etrumadenant; Drug: nanoparticle albumin-bound paclitaxel (NP)
- Dose Escalation-Arm C (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period.
  Interventions: Drug: Etrumadenant; Drug: IPI-549; Drug: Pegylated liposomal doxorubicin (PLD)
- Dose Expansion-TNBC-Arm 1 (Experimental): The dose given will be determined from the dose escalation part (Arm A).
  Interventions: Drug: Etrumadenant; Drug: Pegylated liposomal doxorubicin (PLD)
- Dose Expansion-Ovarian Cancer-Arm 2 (Experimental): The dose given will be determined from the dose escalation part (Arm A).
  Interventions: Drug: Etrumadenant; Drug: Pegylated liposomal doxorubicin (PLD)
- Dose Expansion-TNBC-Arm 3 (Experimental): The dose given will be determined from the dose escalation part (Arm B). .
  Interventions: Drug: Etrumadenant; Drug: nanoparticle albumin-bound paclitaxel (NP)
- Dose Expansion-TNBC-Arm 4 (Experimental): The dose expansion will be determined from the dose escalation part (Arm C).
  Interventions: Drug: Etrumadenant; Drug: IPI-549; Drug: Pegylated liposomal doxorubicin (PLD)

INTERVENTIONS:
Drug: Etrumadenant — Etrumadenant is an A2aR and A2bR antagonist for oral use
  Other Names: AB928
Drug: IPI-549 — IPI-549 is a phosphoinositide-3-kinase-gamma inhibitor for oral use
  Arms: Dose Escalation-Arm C; Dose Expansion-TNBC-Arm 4
Drug: Pegylated liposomal doxorubicin (PLD) — Doxil is an anthracycline topoisomerase II inhibitor that is encapsulated in liposomes for intravenous (IV) use
  Arms: Dose Escalation-Arm A; Dose Escalation-Arm C; Dose Expansion-Ovarian Cancer-Arm 2; Dose Expansion-TNBC-Arm 1; Dose Expansion-TNBC-Arm 4
Drug: nanoparticle albumin-bound paclitaxel (NP) — NP is a microtubule inhibitor for intravenous (IV) use
  Arms: Dose Escalation-Arm B; Dose Expansion-TNBC-Arm 3

SUMMARY:
This is a Phase 1/1b, open-label, dose-escalation, and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and clinical activity of etrumadenant (AB928) in combination with pegylated liposomal doxorubicin (PLD) with or without IPI-549 in participants with advanced metastatic triple-negative breast cancer (TNBC) or ovarian cancer, and etrumadenant in combination with nanoparticle albumin-bound-paclitaxel (NP) in participants with advanced metastatic TNBC.

DETAILED DESCRIPTION:
In the dose escalation phase, the following will be assessed:

* Arm A: escalating doses of etrumadenant in combination with PLD at standard doses will be assessed in participants with advanced metastatic triple-negative breast cancer or ovarian cancer. Eligible participants will receive oral administration of etrumadenant as well as intravenous (IV) infusion of PLD. The recommended dose (RDE) for expansion Arms 1 and 2 and escalation Arm C will be determined upon completion of this dose escalation arm.
* Arm B: escalating doses of etrumadenant in combination with the NP at standard doses will also be assessed in participants with advanced metastatic TNBC. Eligible participants will receive oral administration of etrumadenant as well as NP infusion. The RDE of etrumadenant will be determined upon completion of this dose escalation arm.
* Arm C: escalating doses of IPI-549 in combination with the RDE of etrumadenant (from Arm A) and PLD at standard doses will be assessed in participants with advanced metastatic TNBC or ovarian cancer. Eligible participants will receive oral administration of both etrumadenant and IPI-549 as well as IV infusion of PLD. The RDE of IPI-549 for expansion Arm 4 will be determined upon completion of this dose escalation arm.

In the dose expansion phase, the following will be assessed:

* Arms 1 and 2: Etrumadenant at the RDE in combination with PLD at standard doses may be assessed in participants with advanced metastatic TNBC or ovarian cancer.
* Arm 3: Etrumadenant at the RDE in combination with NP at standard doses may be assessed in participants with advanced metastatic TNBC.
* Arm 4: Etrumadenant and IPI-549 at the RDE in combination with PLD at standard doses may be assessed in participants with advanced metastatic TNBC.

Overall duration of treatment will depend on how well the treatment is tolerated. Treatment may continue until unacceptable toxicity or progressive disease or other reasons specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, 18 years or older
* Measurable disease per radiographic evaluation
* Performance status 0 or 1
* Available archival tissue sample (within 2 years) or a fresh tumor biopsy may be required
* Adequate organ, cardiac, and bone marrow function
* Dose escalation

  * Participants with breast cancer:

    * Locally advanced or metastatic triple negative breast cancer (ER-negative, PgR-negative, and HER2-negative according to ASCO/CAP guidelines) with disease progression
    * No available alternative or curative therapy
    * Participants may have received any number of prior therapies for advanced/recurrent and progressive disease
  * Participants with ovarian cancer:

    * Locally advanced or metastatic ovarian cancer with disease progression
    * No available alternative or curative therapy
    * Participants may have received any number of prior therapies for advanced/recurrent and progressive disease
* Dose expansion

  * Participants with breast cancer:

    * Locally advanced or metastatic triple negative breast cancer (ER-negative, PgR-negative, and HER2-negative according to ASCO/CAP guidelines)
    * Disease progression after no more than 3 prior lines of therapy
  * Participants with ovarian cancer:

    * Locally advanced or metastatic ovarian cancer that is platinum-resistant
    * Disease progression after no more than 3 prior lines of therapy

Exclusion Criteria:

* Received a live, attenuated vaccine within 4 weeks prior to first study treatment
* Prior anticancer treatment including approved agents, systemic radiotherapy, or investigational therapy within 4 weeks prior first study treatment
* Cancer other than the disease under study within 2 years prior to study entry, except for some cancers with a low risk of spreading like non-melanoma skin cancers
* Inability to swallow oral medications
* Participant is breastfeeding, pregnant, or expects to become pregnant during the study
* Active autoimmune disease or documented history of autoimmune disease within 2 years prior to first study treatment
* History of peptic ulcer or stomach bleeding within 6 months prior to first study treatment
* Use of drugs contraindicated by the protocol within 4 weeks prior to and during study treatment
* Prior treatment with drugs that suppress the immune system within 2 weeks prior to first study treatment
* Presence of metastases in the brain or cancer spreading into the cerebrospinal fluid - CSF (leptomeningeal disease)
* HIV, Hepatitis B, and C test results negative prior to first study treatment
* Major surgery within 4 weeks prior to first study treatment
* Participants who have previously received maximum cumulative lifetime anthracycline dosage or baseline ejection fraction <50% (on heart echography)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first dose date to 30 days after the last dose (Approximately 1 year)
Incidence of dose-limiting toxicities (DLTs) during the dose escalation phase | From first dose date to 28 days after the first dose

SECONDARY OUTCOMES:
Plasma concentration of etrumadenant | Recorded at baseline (prior to first dose), during the first 4 cycles of treatment (4 months) and at the end of treatment (i.e. in total approximately 5 months)
Plasma concentration of IPI-549 | Recorded at baseline (prior to first dose), during the first 4 cycles of treatment (4 months) and at the end of treatment (i.e. in total approximately 5 months)
Percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR), as determined by Investigator according to Response Evaluation in Solid Tumors (RECIST) v 1.1 | From study enrollment until participation discontinuation, first occurrence of progressive disease or death from any cause, whichever occurs first (approximately 3-5 years)
Percentage of participants with Disease Control (complete response, partial response, or stable disease) for > 6 months as determined by RECIST v1.1 | From study enrollment until disease progression or loss of clinical benefit (up to approximately 3-5 years)
Duration of Response as determined by the Investigator according to RECIST v1.1 | From the date of the first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
Progression Free Survival (PFS) as determined by the Investigator according to RECIST v1.1 | From start of the treatment up to first occurrence of progressive disease or death from any cause, whichever occurs first (up to approximately 3-5 years)
Overall Survival (OS) as determined by the Investigator according to RECIST v1.1 | From start of treatment up to death from any cause (up to approximately 3-5 years)
Percentage of etrumadenant target inhibition in peripheral blood | Cycle 1 Day 1 through Cycle 4 Day 1 (4 months) and at the end of treatment (in total approximately 5 months)
Immunophenotyping activity in select immune subsets for etrumadenant and IPI-549 in peripheral blood | Cycle 1 Day 1 through Cycle 4 Day 1 (4 months) and at the end of treatment (in total approximately 5 months).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (27):
- United States (20):
  - Scottsdale Healthcare Hospitals dba Honor Health Research Institute, Scottsdale, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Rocky Mountain Cancer Centers (Aurora), Aurora, Colorado
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Maryland Oncology Hematology, PA, Rockville, Maryland
  - HealthPartners Institute Cancer Care Center, Saint Paul, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology, P.A. - Austin (Midtown), Austin, Texas
  - Texas Oncology, P.A. - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology, P.A. - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology, P.A. - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Medical Oncology Associates dba Summit Cancer Centers, Spokane, Washington
  - MultiCare Regional Cancer Center, Tacoma, Washington
- Australia (7):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - St. George Private Hospital, Kogarah, New South Wales
  - Macquarie University, Macquarie, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-2 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=ARC-2